CLINICAL TRIAL: NCT03593070
Title: Dementia Caregiver Chronic Grief Management: A Live Online Video Intervention
Acronym: CGMI-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AG056393-01A1 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Grief; Dementia Family Caregivers
Keywords: online group intervention

STUDY DESIGN:
Intervention Model Description: Study Design The study is a Stage I longitudinal randomized clinical trial. Alzheimer's disease or a related dementia (ADRD) caregivers whose family members are in long-term care facilities will be recruited, screened for inclusion criteria, and will be randomly assigned to either Chronic Grief Management Intervention-Video (CGMI-V) or a Minimal Treatment (MT) condition. Caregivers in the CGMI-V condition will participate in eight weekly professionally led, real-time, live-streaming video online group sessions. Those caregivers in the MT condition will receive written information materials about late-stage ADRD at baseline. For both conditions, data will be collected at baseline (pre-intervention), 8 weeks (immediately post-intervention) for intervention effects, and 24 week post baseline for maintenance effects. The design for this study was chosen to avoid the type of group clustering or contamination that would be engendered by the use of a randomized cluster design.
Who Masked: Outcomes Assessor
Masking Description: Data Collectors will be blinded to the intervention. Study participants will be asked to not disclose their treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGMI-V (Experimental): Caregivers in the Chronic Grief Management Intervention-Video (CGMI-V) condition will participate in eight weekly professionally led, real-time, live-streaming video online group sessions.
  Interventions: Behavioral: Chronic Grief Management Intervention-Video
- Minimal Treatment (MT) (No Intervention): Those caregivers in the MT condition will receive written information materials about late-stage Alzheimer's disease or a related dementia at baseline.

INTERVENTIONS:
Behavioral: Chronic Grief Management Intervention-Video — The CGMI-V participant manual will be provided to participants either mailed or emailed. We will mail hard copies of the manual to caregivers who prefer them over the e-format. The technology assistant will review with each participant the use of technology Cisco WebEx and iPads) via e-mailed step-by-step written instructions and over-the-phone conferencing. Group sessions will take place using WebEx (an internet platform providing video connection) and iPads, at mutually agreed-upon times and days of the week. All group sessions will be audio and video-recorded for fidelity purposes, with caregivers' approval documented in the informed consent. The interventionists will label each recorded meeting group identification number, session number, and date.
  Other Names: CGMI-V
  Arms: CGMI-V

SUMMARY:
The exponential rise in the number of persons diagnosed with Alzheimer's disease and related dementias (ADRD) places a heavy burden on family caregivers. The caregiver role that extends well beyond the placement of the care recipient in long-term care is associated with chronic grief, depressive and anxiety symptoms, dissatisfaction with care, and conflict with long-term care facility staff. This study will test the effects of a cost effective chronic grief management intervention to be delivered using an online platform (Adobe Connect) and iPads. The study aims to decrease dementia caregivers' chronic grief, depressive and anxiety symptoms, and to improve their positive states of mind; to improve satisfaction with care post-placement and to attenuate caregivers' conflict with facility staff.

DETAILED DESCRIPTION:
Evidence indicates that Alzheimer's disease or a related dementia (ADRD) family caregivers suffer long-term mental and physical health effects that place them at risk for premature death. They do not relinquish their role after placing a family member with Alzheimer's disease or a related dementia (ADRD) in long-term care. In fact, these caregivers experience increased symptoms of depression, symptoms of anxiety, and chronic grief post-placement. In the long-term care (LTC) environment, caregivers' chronic grief is exacerbated by their lack of knowledge about late-stage Alzheimer's disease or a related dementia (ADRD) and their sense of loss, guilt, and role captivity. Interventions targeting improvement of ADRD caregivers' mental health have focused overwhelmingly on in-home care. We tested a Chronic Grief Management Intervention (CGMI) with ADRD caregivers in in long-term care and found it feasible (recruitment, retention, and attendance). The Chronic Grief Management Intervention (CGMI) had significant effects on caregiver knowledge and mental health outcomes (heartfelt sadness/longing and guilt; aspects of chronic grief). Although caregivers reported high satisfaction with this intervention, many could not attend the 12 face-to-face group sessions due to the burden of time and competing responsibilities. Therefore, we reduced the number of sessions to 8 and adapted the Chronic Grief Management Intervention to be delivered as a live streaming video, online group intervention; Chronic Grief Management Intervention-Video (CGMI-V), using Adobe Connect (online platform) and iPads. We tested CGMI-V in a single group pilot study for feasibility (recruitment, retention, attendance and technology ease of use) with Alzheimer's disease or a related dementia (ADRD) caregivers post-placement. We obtained 100% retention with high caregiver satisfaction with the intervention and the online technology used to deliver it. Our proposed study, Chronic Grief Management: A Live Streaming Video, Online Intervention (CGMI-V) builds on these results and is guided by a Model of Dementia Caregiver Chronic Grief in the Long-Term Care Setting. The purpose of this study is to test the effects of the 8-week CGMI-V on a caregiver primary outcome (chronic grief); a secondary mental health outcome (symptoms of depression, symptoms of anxiety, and positive states of mind) and a secondary facility-related outcome (caregiver satisfaction with care and conflict with facility staff) related to a minimal treatment (MT) control group. We propose to test the group-based Chronic Grief Management Intervention-Video (CGMI-V) in a Stage I longitudinal, randomized clinical trial. 144 Alzheimer's disease or a related dementia (ADRD) caregivers whose family members reside in one of the participating long-term care facilities will be randomly assigned to either CGMI-V or MT condition. Caregivers in the Chronic Grief Management Intervention-Video (CGMI-V) condition will participate in 8 weekly live streaming video, online group sessions. Caregivers in the minimal treatment (MT) condition will receive written information about late-stage ADRD at baseline. For both conditions, data will be collected at baseline, 8 weeks (immediately post-intervention) and then at 24 weeks post-baseline, using measures of caregiver grief: Marwit-Meuser Caregiver Grief Inventory(MM-CGI); depressive symptoms: Center for Epidemiological Studies Depression Scale (CES-D); anxiety symptoms: Stait-Trait Anxiety Inventory (STAI); positive states of mind: Positive States of Mind Scale (POSMS); satisfaction with care: Family Perception of Care Tool (FPCT); conflict with facility staff: Family Perception of Caregiving Role (FPCR subscale), knowledge of Alzheimer's disease: Family Knowledge of Alzheimer's Test (FKAT), loss, guilt and role captivity (FPCR subscales). Specific aims are to: 1) Establish effect sizes of the Chronic Grief Management Intervention-Video (CGMI-V) condition and Minimal Treatment (MT) control condition on changes in caregiver chronic grief. 2) Establish effect sizes of the CGMI-V and Minimal Treatment (MT) control condition on changes in caregiver symptoms of depression and anxiety and on positive states of mind. 3) Establish effect sizes of the CGMI-V condition and the Minimal Treatment (MT) control condition on changes in caregiver satisfaction with care provided in the facility and conflict with staff, and 4) Explore mechanisms of intervention impact on all caregiver outcomes. Our long-term objective is to develop a chronic grief treatment modality that will be adopted in long-term care facilities as part of routine support for Alzheimer's disease or a related dementia caregivers post-placement. This in turn will impact public mental health for this growing segment of the population.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Identified as family member, fictive kin (self-identified family member), or partner of care recipient at any time post permanent placement of care in long-term care facility (LTCF)
* Care recipient has a documented ADRD diagnosis and resides in any type of unit in a LTCF
* Possessing self-reported basic computer literacy and in-home internet access
* Able to speak, read, and write English
* Not currently attending another ADRD caregiver grief management group
* Experiencing high to moderate levels of grief per screening with the Marwit-Meuser Caregiver Grief Inventory-Short Form (MMCGI-SF) (70 and above); and/or
* Experiencing high levels of depressive symptoms per screening with Patient Health Questionnaire-9 (PHQ-9) (scores 10 and above)

Exclusion Criteria:

* Non English speaker, reader, writer
* Scoring under the cut off points on the MM-CGI-SF and the PHQ-9
* Reporting no basic computer literacy; no internet access

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olimpia Paun, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Paun O, Loukissa D, Chirica MG, Nowell HM 3rd. Loss and Grief in the Context of Dementia Caregiving. J Psychosoc Nurs Ment Health Serv. 2022 Oct;60(10):7-10. doi: 10.3928/02793695-20220909-01. Epub 2022 Oct 1. PMID 36179053
- See also: DOI: 10.3928/02793695-20220909-01 — https://pubmed.ncbi.nlm.nih.gov/36179053/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGMI-V | Minimal Treatment (MT)
Started | 50 | 49
Completed | 49 | 48
Not Completed | 1 | 1
Not completed — administrative withdrawal | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic characteristics of sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | CGMI-V | Minimal Treatment (MT) | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.9) | 58.5 (11.2) | 60.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 44 | 43 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 42 | 33 | 75
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Marwit Meuser Caregiver Grief Inventory (MM-CGI) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 50 to 250; higher scores represent higher levels of grief.
  units on a scale | 152.16 (29.90) | 164.46 (34.27) | 158.24 (32.56)

OUTCOME MEASURES:

1. Primary Outcome: Marwit-Meuser Caregiver Grief Inventory (MM-CGI)
Description: Marwit-Meuser Caregiver Grief Inventory (MM-CGI). Scores range from 50 to 250; higher scores represent higher levels of grief.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Population: Study data for 97 participants were analyzed, to determine the mean difference in CGMI-V scores from baseline to 24 weeks. The CGMI-V group was analyzed on an intent to treat (ITT) basis. At baseline, 49 participants were assigned to the CGMI-V group, of whom 44 provided data at Week 8 and 47 provided data at week 24. At baseline, 48 participants were assigned to the MT condition, of whom 45 provided data at Week 8 and 43 provided data at week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 12.75 (9.01) | 11.04 (7.81)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in total scores for the MM-CGI from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.646, Standard Deviation 0.622

2. Secondary Outcome: Change in Depressive Symptoms
Description: Center for Epidemiological Studies Depression Scale (CES-D). The CES-D was assessed with 20-items, where responses are based on a four-point frequency rating (0 = rarely or none of the time to 3 = all of the time), with a possible range of 0 to 60. Larger scores represent more depressive symptoms, lower scores represent fewer symptoms.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 6.45 (4.56) | 0.87 (0.62)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Analyses compared changes in total scores for the CESD from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); Test type: Other; p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.444, Standard Deviation 0.105

3. Secondary Outcome: Change in Anxiety Symptoms
Description: State-Trait Anxiety Inventory (STAI) was used to represent anxiety symptoms. The (STAI) includes 20 questions, with responses based on a scale of 1 to 4 (1 = almost never to 4 = almost always). Numeric responses to these questions are summed to produce an inventory score, with a possible range of 20-80, where higher scores indicate greater anxiety, and lower scores indicate less anxiety.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 5.77 (4.08) | 0.86 (0.61)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in total State Trait Anxiety Inventory (STAI) scores from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.514, Standard Deviation 0.102

4. Secondary Outcome: Change in Positive States of Mind
Description: Positive States of Mind Scale (PSOMS) was used to assess the extent to which caregivers were able to achieve six positive states of mind in the previous seven days. PSOM is based on 6 questions that are scored 0-4 and which are summed to produce scale scores that range from 0-24. Lower scores represent difficulty achieving positive states of mind in the past 7 days, higher scores indicate less difficulty achieving positive states of mind.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 1.60 (1.13) | 0.11 (0.08)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in total positive state of mind scale (PSOMS) scores from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.653, Standard Deviation 0.093

5. Secondary Outcome: Change in Conflict With Facility Staff
Description: Conflict with facility staff was assessed with a subscale of 10 questions collected in the Family Perception of Caregiving Role (FPCR) tool. Scores on these 10 questions ranged from 1 (strongly disagree) to 7 (strongly agree). Response values associated with conflict subscale items were summed to produce total conflict scores ranging from 10-70. Lower scores indicate less conflict with facility staff, higher scores indicate more conflict with facility staff.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 3.83 (2.71) | 3.75 (2.65)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in conflict scores (based on FPCR) from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.609, Standard Deviation 0.070

6. Secondary Outcome: Change in Satisfaction With Care
Description: The Family Perception of Care Tool (FPCT) is comprised of 51 questions with 7-point likert-type responses where 1=strongly agree and 7=strongly disagree. When summed to create a total FPCT score, values ranged from 51-357. Higher scores in the FPCT represent more positive feelings towards staff whereas lower scores represent more negative feelings.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 2.98 (2.11) | 9.73 (6.88)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in total scores for satisfaction with care measure (FPCT) from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.731, Standard Deviation 0.074

7. Other Pre Specified Outcome: Change in Knowledge of Alzheimer's Disease
Description: Family Knowledge of Alzheimer's Tool (FKAT) captures what a family caregiver knows about the disease process, how the care recipient is behaving, and how the long-term care facility (LTCF) is caring for him or her. Responses are based on a true/false scale, with scores ranging from 0 to 22 correct answers; larger scores indicate greater knowledge about AD, lower scores indicate less knowledge about AD.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 0.29 (0.21) | 0.39 (0.28)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Test type: Other — Analyses compared changes in total Family Knowledge of Alzheimer's Test (FKAT) scores from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT); p = 0.001, Regression, Linear — A priori alpha=0.05; Slope = 0.687, Standard Deviation 0.084

8. Other Pre Specified Outcome: Change in Caregiver Sense of Loss, Guilt, and Role Captivity
Description: The Revised Family Perceptions of Caregiving Role (FPCR) instrument includes subscales for Loss, Guilt, Role Captivity, and Conflict. Using revised subscales for Loss (7 items), Guilt (5 items), and Role Captivity (7 items), a total score for each subscale was calculated by summing numerical responses to the related questions. The scale ranges were:
  Loss (7-49), Guilt (5-35), Role Captivity (7-49).
  Each of the subscales (Sense of Loss, Guilt, and Role Captivity) were then summed to provide a Total score for FPCR, scores of which ranged from 19-133.
  For each of the subscales and the Total, higher scores represent more negative perceptions of the Caregiving Role, lower scores represent improved perceptions of the Caregiving Role.
Time Frame: Measured at Baseline, 8 weeks, and 24 weeks, Baseline to 24 weeks reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGMI-V | Minimal Treatment (MT)
Number analyzed (Participants) | 49 | 48
units on a scale | 3.84 (2.72) | 4.58 (3.24)
Statistical Analysis 1: Comparison: CGMI-V vs Minimal Treatment (MT); Analyses compared changes in caregiver sense of loss, guilt, and role captivity scores from baseline to 24 weeks, for both arms of the intervention (CGMI-V and MT). This measure uses 51 items of the FPCR measure; Test type: Other; p = 0.001, Regression, Linear — A prior alpha=0.05; Slope = 0.527, Standard Deviation 0.088

ADVERSE EVENTS:
Time Frame: Participants were assessed for depressive symptoms at Baseline, 8 weeks, and 24 weeks.
Description: For the purposes of this study, adverse events were considered participants scoring above a 16 on the CES-D (Center for Epidemiological Studies Depression Scale) at assessment points (8 weeks and 24 weeks). All participants scoring above 16 on the CES-D were contacted by the study PI, who evaluated the severity of depressive symptoms (mild, moderate, severe). None of the participants' elevated CES-D levels were determined to be related to study participation.
Arm/Group | CGMI-V | Minimal Treatment (MT)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

LIMITATIONS AND CAVEATS:
One limitation is that this trial was conducted while dementia family caregivers and long-term care facilities were severely affected by the COVID-19 pandemic. Study recruitment was impacted- the final sample was less than planned (97 v. 144 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03593070/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT03593070/ICF_000.pdf